CLINICAL TRIAL: NCT07089160
Title: Decision Fatigue Among Anesthesiologists: The Relationship Between Cognitive Load and Emotional Exhaustion
Brief Title: Decision Fatigue and Emotional Exhaustion Among Anesthesiologists
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Other Study IDs: HASEKİ KARAR
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Online Survey (Decision Fatigue Scale and Emotional Exhaustion Scale) — Participants will complete an online survey including demographic questions, the Decision Fatigue Scale (DFS), and the Emotional Exhaustion subscale of the Maslach Burnout Inventory.

SUMMARY:
This study aims to evaluate the level of decision fatigue among anesthesiologists actively practicing in clinical settings in Turkey and to examine its relationship with emotional exhaustion. Participants will complete an online survey including demographic information, the Decision Fatigue Scale (DFS), and the Emotional Exhaustion subscale of the Maslach Burnout Inventory. The study will explore associations between decision fatigue scores and demographic or professional variables, as well as correlations with emotional exhaustion levels. Data will be collected anonymously and analyzed to identify factors contributing to cognitive load and burnout among anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* Actively practicing anesthesiologists (specialists or residents) in Turkey.
* Age 24 years or older.
* Voluntarily provides informed consent through the online form.
* Completes the online survey in full.

Exclusion Criteria:

* Health care professionals not working in the field of anesthesiology.
* Individuals who do not provide informed consent through the online form.
* Participants who submit incomplete surveys or provide patterned/invalid responses that compromise data quality.
* Physicians currently in administrative positions who are not actively involved in clinical decision-making processes.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Actively practicing anesthesiology specialists and residents in Turkey, aged 24 years or older, who voluntarily complete an online survey.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Decision Fatigue Score measured by the Decision Fatigue Scale (DFS) | three minutes
  The primary outcome is the total score obtained from the Decision Fatigue Scale (DFS). Higher scores indicate greater decision fatigue. The scale will be administered once through an online questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Result] Pignatiello GA, Martin RJ, Hickman RL Jr. Decision fatigue: A conceptual analysis. J Health Psychol. 2020 Jan;25(1):123-135. doi: 10.1177/1359105318763510. Epub 2018 Mar 23. PMID 29569950
- [Result] Grignoli N, Manoni G, Gianini J, Schulz P, Gabutti L, Petrocchi S. Clinical decision fatigue: a systematic and scoping review with meta-synthesis. Fam Med Community Health. 2025 Feb 8;13(1):e003033. doi: 10.1136/fmch-2024-003033. PMID 39922690